CLINICAL TRIAL: NCT05308524
Title: Role of Disease Severity Scoring Systems in Predicting Mortality covid19 Pts in AUH
Brief Title: Scoring Systems covid19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebtesam Mohamed Thabet, resident doctor, Assiut University
Other Study IDs: ICU scoring system in covid19
Record Dates: First submitted 2022-03-31; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: ICU Scoring System in Covid 19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ICU scoring system in covid 19 — The intensive care unit (ICU) at Assiut University Hospital, which is supervised by the staff members of the Chest Diseases Department and designated to deal with critically ill Covid 19 patients.

SUMMARY:
In this study, we planned to investigate the role and determine the predictive performance of both APACHE II and SAPS II scoring systems and compare them in COVID-19 patients admitted to the intensive care unit of Assiut University Hospital.

DETAILED DESCRIPTION:
Since the start of the coronavirus disease 2019 (COVID-19) pandemic, intensive care units (ICUs) worldwide have struggled to treat affected patients who require a completely different approach to treatment than other patients

* [1]* .This study aims to evaluate the efficacy of single dose analgesia in combination with local anaesthesia to control pain during TUS guided procedures. It also aims to assess the effect of its use on procedure performance time and rate of complications occurrence compared to local anaesthesia alone.Although many severe cases are admitted to ICUs, it is unknown whether the conventional disease-severity scoring systems that were developed for ICU patients can be applied to patients with COVID-19.Several recent studies have used Acute Physiology and Chronic Health Evaluation (APACHE) and Simplified Acute Physiology Score (SAPS) to provide information on the clinical severity of COVID-19
* [2-4]*. However, very few reports have examined their validity of applying them to patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:•

* • This study will be conducted on laboratory-confirmed COVID-19 patients who will be transferred to the intensive care unit of Assiut University Hospital

Exclusion Criteria:

* Patients would be excluded from this study if they died or were discharged from the intensive care unit prior collection of data required for both the APACHE II and SAPS II scoring systems, if they were discharged before their outcomes were determined and if we could not obtain consent from them or their companions to participate in this study. All patients involved will be subjected to a full history with special stress on age, gender, special habits, and associated diseases. Information such as the patient's need for ventilatory support as well as the length of ICU stay will be entered. Also, the laboratory results and Imaging findings will be registered. Scores of APACHE II and SAPS II were calculated as illustrated in the previously published works *[5,6]* .Patients will be followed up until their outcome was determined.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sample size was calculated using Epi- Info7. Based on previous studies the mortality rate of Covid-19 ICU admitted patients varies between countries, in low resources sittings the mortality rate was around 50% *[7 ]*. With a confidence limits of 10% and a confidence level of 90% the minimum number of patients required for this study is 70 patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
ICU scoring system in covid 19 | Baseline
  SAPS ,APACHE ICU scoring system in covid 19

REFERENCES:
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Michard F, Vieillard-Baron A. Critically ill patients with COVID-19: are they hemodynamically unstable and do we know why? Intensive Care Med. 2021 Feb;47(2):254-255. doi: 10.1007/s00134-020-06238-5. Epub 2020 Sep 10. No abstract available. PMID 32910203